CLINICAL TRIAL: NCT00138606
Title: Extension to a Study on the Efficacy and Safety of Vildagliptin in Combination With Insulin in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLAF237A2311E1
Record Dates: First submitted 2005-08-27; First posted 2005-08-30 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 diabetes; vildagliptin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin

INTERVENTIONS:
Drug: vildagliptin

SUMMARY:
Many people with type 2 diabetes cannot maintain their target blood glucose levels on a single therapy. This is a 28-week extension to a study to assess the safety and effectiveness of vildagliptin, an unapproved drug, in lowering overall blood glucose levels when added to insulin in people with type 2 diabetes who are not at target blood glucose levels on insulin alone. The purpose of the extension study is to gather data on the long-term safety and effectiveness of vildagliptin in people with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Only patients successfully completing study CLAF237A2311 are eligible
* Written informed consent
* Ability to comply with all study requirements

Exclusion Criteria:

* Premature discontinuation from CLAF237A2311
* Other protocol-defined exclusion criteria may apply

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2005-01; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Safety of vildagliptin in combination with insulin during 52 weeks of treatment
Change from baseline in HbA1c at 52 weeks

SECONDARY OUTCOMES:
Change in HbA1c between 24 weeks and 52 weeks
Change in fasting plasma glucose between 24 weeks and 52 weeks
Change from baseline in fasting plasma glucose at 52 weeks
Change from baseline in mean daily insulin dose at 52 weeks
Change from baseline in mean daily number of insulin injections at 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States
- Novartis Investigative Site, Investigative Centers, Germany

REFERENCES:
- [Result] Fonseca V, Baron M, Shao Q, Dejager S. Sustained efficacy and reduced hypoglycemia during one year of treatment with vildagliptin added to insulin in patients with type 2 diabetes mellitus. Horm Metab Res. 2008 Jun;40(6):427-30. doi: 10.1055/s-2008-1058090. Epub 2008 Mar 11. No abstract available. PMID 18401832